CLINICAL TRIAL: NCT00181220
Title: Valproic Acid in the Induction of EBV Lytic Cycle Antigen Expression in Nasopharyngeal Carcinoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left JHU and is not able to be reached for updates
Sponsor: Johns Hopkins University (Other)
Collaborators: National University Hospital of Singapore (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Valproic Acid NPC
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2019-05

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Valproic Acid

INTERVENTIONS:
Drug: valproic acid

SUMMARY:
The proposed study will test the safety and efficacy of sodium valproate in the induction of Epstein-Barr virus (EBV) lytic cycle antigen expression in tumor tissue of patients undergoing primary therapy for nasopharyngeal carcinoma. Up to 20 patients will be given valproic acid for 2 weeks. The primary surrogate endpoint for efficacy will be expression of EBV lytic antigens by immunohistochemistry in tumor tissue. Biopsies of primary tumor will be taken after 2 weeks with achievement of a therapeutic concentration of valproate. Expression of immunodominant EBV latency antigens in tumor tissue, EBV viral load by real time PCR, and valproate levels will be measured. Adverse events associated with valproate in NPC patients will be described.

ELIGIBILITY:
Inclusion Criteria:

All subjects must fulfill the following criteria to be eligible for study admission:

* Subjects are of age 18 years and above
* Biopsy proven nasopharyngeal carcinoma - WHO type 3
* Must have tumor which is accessible to biopsy
* For patients with disease localized to the PNS, the lesion must be visualized by endoscopy
* Subjects with metastatic disease with disease accessible to biopsy in the PNS if they are deemed by their treating physicians not to require treatment for at least two weeks.
* An ECOG performance status of 0-2
* For sexually active women of child-bearing potential, negative pregnancy test within 14 days of enrolling on trial
* Must be able to give informed consent

Exclusion Criteria:

* For patients with localized NPC, PNS lesions that cannot be visualized by endoscopy
* Patients with disease inaccessible to biopsy
* History of anaphylaxis after exposure to valproic acid
* Hepatic dysfunction as defined by total bilirubin 1.0x upper limit of normal. AST (SGOT) and ALT (SGPT) 3x upper limit of normal
* Hemoglobin 8g/dl, Absolute neutrophil count 1500 cells/mm, and Platelet count 100,000 /mm
* Creatinine 3x upper limit of normal
* PT/PTT blood test result not within normal range
* Patients who require treatment with an anticonvulsant besides valproic acid during the course of valproate prescribed by the protocol
* ECOG Performance status 3-4
* Patients who are pregnant or breast feeding (Sexually active women of childbearing potential must use contraception during course of therapy and within 4 weeks of completion of trial)
* Participation in another clinical trial involving therapeutic intervention within 4 weeks of enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-04; Study Completion 2006-09

PRIMARY OUTCOMES:
expression of EBV lytic cycle antigens in NPC tumor tissue. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wen-son Hsieh, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkin Singapore International Medical Center, Singapore, Singapore